CLINICAL TRIAL: NCT00290849
Title: European Registry of Consecutive Patients Undergoing PCI Evaluating the Use of the Thrombin-specific Anticoagulant Bivalirudin With Focus on Patient Selection, Convenience and Safety Aspects.
Brief Title: ImproveR International (BI-001-IM)
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Clinical Trial Operations
Other Study IDs: BI-001-IM
Record Dates: First submitted 2005-12-14; First posted 2006-02-13 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2010-04

CONDITIONS: Thrombin-specific Anticoagulant Bivalirudin During Percutaneous Coronary Intervention (PCI)
MeSH Terms: interventions — bivalirudin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bivalirudin

SUMMARY:
The objectives of this registry are to assess the use of the thrombin-specific anticoagulant bivalirudin during percutaneous coronary intervention (PCI) in a real life setting. In particular, data will be collected to analyze experiences of bivalirudin use in respect to the following objectives;

* examine the aspects of safety and effectiveness of bivalirudin
* gain experience regarding the characteristics of patients in bivalirudin treatment
* evaluate the handling of bivalirudin and its practicality

ELIGIBILITY:
Inclusion Criteria:

> 18 years, undergoing planned or urgent PCI with the intention to use bivalirudin as anticoagulant, written informed concent to entry of data information registry.

Exclusion Criteria:

None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 4000
Dates: Start 2005-03; Primary Completion 2006-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To assess the use of the thrombin-specific anticoagulant bivalirudin during percutaneous coronary intervention (PCI) in a real life setting. In particular, data will be collected to analyze experiences of bivalirudin use in respect to the following;
•examine the aspects of safety and effectiveness of bivalirudin
•gain experience regarding the characteristics of patients in bivalirudin treatment
•evaluate the handling of bivalirudin and its practicality.

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquaters
Locations (1):
- Nycomed, Roskilde, Denmark